CLINICAL TRIAL: NCT07292246
Title: A Prospective CohorT Study of HandX - Assisted ENdoscopic MAstectomy: Feasibility and Safety (ATHENA I Study)
Acronym: ATHENA I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vasileios Kalles (Other)
Responsible Party: Sponsor-Investigator, Vasileios Kalles, Vasileios Kalles MD, MSc, PhD, FEBS, Consultant Breast & General Surgeon, Director of Mediterraneo Breast Clinic, Mediterraneo Hospital
Organization: Mediterraneo Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 516
Record Dates: First submitted 2025-11-25; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; BRCA 1 Gene Mutation; BRCA 2 Gene Mutation; Hereditary Breast Carcinoma; Breast Neoplasms; DCIS; Germline Mutation Abnormality; Early Breast Cancer
Keywords: breast cancer; mastectomy; endoscopic; robotic; handx; nipple-sparing mastectomy
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer, Familial; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HandX-assisted endoscopic nipple sparing mastectomy (Experimental): Patient cohort undergoing endoscopic nipple sparing mastectomy with use of HandX.
  Interventions: Procedure: Endoscopic nipple sparing mastectomy; Device: HandX endoscopic instrument

INTERVENTIONS:
Procedure: Endoscopic nipple sparing mastectomy — A minimally invasive nipple-sparing mastectomy performed through a single lateral mammary fold incision using endoscopic visualization and CO₂ insufflation. Breast tissue is dissected from the skin envelope and nipple-areola complex, and immediate implant-based reconstruction is performed according to standard practice. The HandX device is used for articulating endoscopic dissection.
Device: HandX endoscopic instrument — A handheld articulating endoscopic instrument used to assist with endoscopic dissection during nipple-sparing mastectomy. The HandX device provides wrist-like articulation, motion scaling, and ergonomic control during minimally invasive surgery.

SUMMARY:
This study aims to learn whether a handheld robotic device, called the HandX, can help surgeons safely perform a minimally invasive nipple-sparing mastectomy. This type of mastectomy uses a small incision at the side of the breast to remove breast tissue while keeping the skin and nipple in place. The goal is to lower scarring, improve comfort, and support good cosmetic results after surgery.

Participants in this study will already be planning to have a therapeutic or preventive mastectomy with immediate implant-based reconstruction. All surgeries are done at Mediterraneo Hospital in Greece.

During the operation, surgeons use the HandX device to assist with the endoscopic dissection. Researchers will collect information about how long the surgery takes, whether the planned approach can be completed without switching to open surgery, and whether any surgical complications occur. They will also check healing, infection, and implant-related problems for up to 365 days after surgery. Participants will complete the BREAST-Q questionnaire before surgery and at several times after surgery to share their views on comfort, well-being, and cosmetic outcomes.

About 15 participants will take part. The results will help researchers understand whether this approach is practical and safe, and whether it should be studied further in a larger trial.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm interventional study designed to evaluate the feasibility and surgical safety of HandX-assisted endoscopic nipple-sparing mastectomy with immediate implant-based breast reconstruction. The HandX system is a handheld articulating robotic instrument that provides wrist-like motion, motion scaling, and ergonomic control. Unlike console-based robotic platforms, HandX integrates into standard minimally invasive workflows without the need for a large footprint, dedicated console, or complex docking procedures. Early clinical experience in other surgical specialties suggests that the technology may improve access and ergonomics during dissection while maintaining procedural efficiency. This study investigates its use specifically in endoscopic breast surgery, where instrument articulation and visualization are key technical challenges.

All participants will undergo the mastectomy through a single lateral mammary fold incision. Following tumescent injection and creation of a working space, a single-port device is placed, and CO₂ insufflation is used to establish the operative cavity. The HandX device is then employed for endoscopic dissection of the breast gland from the skin envelope and the nipple-areola complex. Specimen retrieval is performed through the same incision. Reconstruction is completed using implant-based techniques (prepectoral, dual-plane, PU-coated, or subpectoral), according to preoperative planning and standard practice. Axillary procedures (sentinel lymph node biopsy or axillary lymph node dissection) may be performed through the same incision when indicated.

The study focuses on technical feasibility-specifically, the ability to complete the endoscopic mastectomy using the HandX platform without unplanned conversion to an open approach. Technical success is defined in the protocol and includes completion of all key steps of the planned minimally invasive procedure. Adjunct use of standard laparoscopic instruments or minor incision extensions for specimen handling does not constitute conversion, provided that the minimally invasive workflow is preserved.

Safety outcomes include intraoperative complications, 30-day and 90-day postoperative adverse events, surgical site infections assessed according to CDC/NHSN definitions, implant-related complications, and implant loss through one year. Postoperative care follows standardized pathways for implant-based reconstruction, including consistent antibiotic and VTE prophylaxis policies and predefined criteria for drain management. Participants are reviewed at scheduled visits through postoperative day 28, with additional follow-up through day 90 for infection surveillance, and through one year for implant-related outcomes.

Patient-reported outcomes are assessed using the BREAST-Q® Reconstruction Module (Version 2.0), administered preoperatively and at postoperative months 1, 6, and 12. These measures provide data on satisfaction with breasts, psychosocial and sexual well-being, physical well-being of the chest, and satisfaction with aspects of care. Only implant-reconstruction-relevant scales are used.

All data are collected in electronic case report forms, stored securely, and managed in compliance with GDPR and institutional policies. Monitoring is internal due to the single-center pilot nature of the study.

The study plans to accrue up to 20 mastectomy cases, corresponding to approximately 15 participants, as bilateral procedures are counted per breast. The sample size of 20 cases is consistent with recommendations for feasibility studies intended to inform future multicenter comparative trials. Analyses are descriptive. Technical success, complication rates, and patient-reported outcomes will be summarized with confidence intervals. Progression criteria and stopping rules are predefined in the protocol, including thresholds for major complications, device-related serious events, and oncologic or surgical concerns that may warrant pause or termination of the study.

Findings from this pilot study will inform the development of larger controlled trials evaluating the comparative effectiveness, aesthetic outcomes, recovery profiles, and cost implications of HandX-assisted endoscopic mastectomy relative to other surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age ≥ 18 years old
* Indication for therapeutic or prophylactic (risk-reducing) mastectomy for:

  1. early invasive breast cancer (Clinical Stage I-II at diagnosis) undergoing primary surgery
  2. early invasive breast cancer (Clinical Stage I-II at diagnosis) undergoing surgery post systemic (neoadjuvant) therapy with clinical evidence of partial or complete response
  3. ductal carcinoma in situ (DCIS), or
  4. BRCA or other breast cancer - related genetic mutation carriers, or
  5. high risk for development of breast cancer.
* Breast volume: cup sizes A to C as defined by underwear size, expected implant volume <550cc and glandular ptosis not exceeding Grade I Regnault's classification.
* ECOG / WHO Performance Status <2
* Subject with signed and dated informed consent form

Exclusion Criteria:

* Chest wall or skin invasion
* Extended lymph node involvement at diagnosis (cN2)
* Inflammatory breast cancer
* Tumor distance from nipple - areola complex <1cm on imaging studies
* Active smoking/nicotine use within 4 weeks pre-op (combustible tobacco, vaping, nicotine pouches, NRT)
* BMI >35
* High risk patients with severe and poorly controlled co-morbid conditions (including but not limited to diabetes, heart disease, renal failure or liver dysfunction)
* Pregnancy or breastfeeding
* Psychiatric, addictive, or any disorders which compromise the ability to give informed consent for participation in this study
* Subject without signed and dated informed consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Technical success | Intraoperative (Day 0)
  Completion of the planned procedure via the minimally invasive approach without unplanned conversion.
Surgical Safety | Postoperative Day 0-30
  Major (Clavien-Dindo ≥III) complications

SECONDARY OUTCOMES:
Operative Time | Intraoperative (Day 0)
  Total Operative Time
Blood Loss | Intraoperative (Day 0)
  Intraoperative Blood Loss
Length of Stay | From hospitalization to discharge (average 1-3 days)
  Length of hospital stay in days
Complications | Within 30 days after surgery
  30-day complication rate (Clavien-Dindo)
Skin flap necrosis | Within 30 days after surgery
  The presence of skin flap necrosis will be noted during all the visits after the surgery (POD 7, 14, 28).
Nipple Areola Complex ischemia | Within 30 days after surgery
  Nipple-Areola-Complex (NAC) Ischemia noted during all the visits after the surgery (POD 7, 14, 28)
Surgical Site Infection | Within 90 days after surgery
  Number of participants with SSI (CDC/NHSN). Superficial incisional primary (SIP) within 30 days; deep incisional primary (DIP) and organ/space (O/S) within 90 days after the index BRST procedure.
Implant loss | Within 1 year after surgery
  Need to remove the implant for any reason
Short - term Oncologic Adequacy | Within 40 days after surgery
  Negative surgical margins on final pathology-retroareolar (nipple) margin negative and no tumor on ink on any sampled skin-flap or deep margin
PROMs - Aesthetic Outcome | Preoperatively up to 4 weeks, 1 month postoperatively, 6 months postoperatively, 12 months postoperatively
  BREAST-Q© questionnaire Version 2.0 measure the quality of life and satisfaction among patients undergoing breast surgery - Reconstruction module pre and postoperative, higher scores reflect a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Kalles, MD, MSc, PhD, FEBS, Principal Investigator — Mediterraneo Hospital
Locations (1):
- Mediterraneo Hospital, Glyfada, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
"Individual participant data (IPD) will not be shared. This study is a small single-center feasibility trial, and the dataset contains clinical and surgical details that cannot be fully de-identified under GDPR. Summary results will be made available in the ClinicalTrials.gov record after study completion.

REFERENCES:
- [Background] Toesca A, Peradze N, Galimberti V, Manconi A, Intra M, Gentilini O, Sances D, Negri D, Veronesi G, Rietjens M, Zurrida S, Luini A, Veronesi U, Veronesi P. Robotic Nipple-sparing Mastectomy and Immediate Breast Reconstruction With Implant: First Report of Surgical Technique. Ann Surg. 2017 Aug;266(2):e28-e30. doi: 10.1097/SLA.0000000000001397. No abstract available. PMID 28692558
- [Background] Jain Y, Lanjewar R, Shinde RK. Revolutionising Breast Surgery: A Comprehensive Review of Robotic Innovations in Breast Surgery and Reconstruction. Cureus. 2024 Jan 21;16(1):e52695. doi: 10.7759/cureus.52695. eCollection 2024 Jan. PMID 38384645
- [Background] Toesca A, Peradze N, Manconi A, Galimberti V, Intra M, Colleoni M, Bonanni B, Curigliano G, Rietjens M, Viale G, Sacchini V, Veronesi P. Robotic nipple-sparing mastectomy for the treatment of breast cancer: Feasibility and safety study. Breast. 2017 Feb;31:51-56. doi: 10.1016/j.breast.2016.10.009. Epub 2016 Nov 2. PMID 27810700
- [Background] Khan MF, Kearns E, Cahill RA. Clinical Experience of a Smart Articulating Digital Device for Transanal Minimally Invasive Surgery. Dis Colon Rectum. 2023 Dec 1;66(12):e1265-e1268. doi: 10.1097/DCR.0000000000002987. Epub 2023 Sep 25. PMID 37787571
- [Background] Mao R, Gao L, Gang W, Wen L. Literature Review of Handheld Articulating Instruments in Minimally Invasive Surgery. J Laparoendosc Adv Surg Tech A. 2024 Jan;34(1):47-54. doi: 10.1089/lap.2023.0366. Epub 2023 Oct 23. PMID 37870762
- [Background] Cao L, Shenk R, Miller ME, Towe C. Minimally Invasive Mastectomy Could Achieve Non-inferior Oncological Outcome in Appropriately Selected Patients: Propensity Matched Analysis of the National Cancer Database. Am Surg. 2022 Dec;88(12):2893-2898. doi: 10.1177/00031348211011152. Epub 2021 Apr 16. PMID 33861667
- [Background] Mok CW, Lai HW. Evolution of minimal access breast surgery. Gland Surg. 2019 Dec;8(6):784-793. doi: 10.21037/gs.2019.11.16. PMID 32042687